CLINICAL TRIAL: NCT02783430
Title: Evaluation of the Initial Prescription of Ketamine and Milnacipran Forin Depression in Patients With a Progressive Disease
Brief Title: Evaluation of the Initial Prescription of Ketamine and Milnacipran in Depression in Patients With a Progressive Disease
Acronym: KETAPAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014_22; 2014-004361-24 (EudraCT Number); PHRCI_2013 (Other: PHRC Number, DGOS)
Record Dates: First submitted 2016-05-12; First posted 2016-05-26 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Depression
Keywords: Ketamine; Palliative care; Supportive care; Early palliative care; Fast acting antidepressant; End of life care; Cancer; psychological distress; antidepressant; serotonin norepinephrine reuptake inhibitors
MeSH Terms: conditions — Depression; Neoplasms | interventions — Ketamine; Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milnacipran + Ketamine (Experimental): Ketamine 0,5mg/kg single intravenous perfusion during 40 minutes. Milnacipran dosage depending of glomerular filtration rate of patient, during 16 days (doses of 25 or 50 mg or 100mg per day)
  Interventions: Drug: Ketamine; Drug: Milnacipran
- Milnacipran + Placebo (Active Comparator): Placebo single intravenous perfusion during 40 minutes. Milnacipran dosage depending of glomerular filtration rate of patient, during 16 days (doses of 25 or 50 mg or 100mg per day)
  Interventions: Drug: Milnacipran; Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — One single perfusion of 0.5 mg/kg during 40 minutes at the beginning of the inclusion
  Arms: Milnacipran + Ketamine
Drug: Milnacipran — One or two caps per day from the beginning of the inclusion. Milnacipran dosage depending of glomerular filtration rate of patient, during 16 days (doses of 25 or 50 mg or 100mg per day)
Drug: Placebo — One single perfusion during 40 minutes at the beginning of the inclusion
  Arms: Milnacipran + Placebo

SUMMARY:
KetaPal is a placebo-controlled randomized trial designed to demonstrate the antidepressant action of ketamine in palliative care situations. Half of participants will receive Ketamine and Milnacipran in combination, while the other half will receive a Placebo and Milnacipran in combination.

DETAILED DESCRIPTION:
Ketamine, a molecule mainly used as an analgesic in palliative care, turns out to be an excellent fast acting antidepressant. By acting as an NMDA receptor antagonist, its mechanism of action is complementary to classical and long acting antidepressants like Selective Serotonin Reuptake Inhibitors (SSRI). In particular, ketamine is able to boost synaptogenesis in only a few hours whereas long-term prescription of SSRI can stimulate neurogenesis.

The purpose of this study is to evaluate a new therapeutic strategy that could integrate ketamine in the same time than SSRI, to control depression symptoms faster and optimize patient's quality of life complementary to treatments of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient
* Supported by a functional palliative care unit
* Having a severe and progressive disease diagnosed
* Meet the criteria for major depressive disorder as defined by DSM in its version 5
* MADRS > 19 ( moderate to severe)
* No antidepressant treatment or treatment introduced for more than four weeks
* In ability to receive clear information and give consent
* Beneficiary of a social security scheme

Exclusion Criteria:

* upper weight or equal to 100 kg
* ultimate phase (about 24 to 72 hours prior to death)
* unstable patient on cardiovascular diseases, including uncontrolled hypertension
* severe renal impairment (renal clearance less than 15 ml / min)
* psychiatric comorbidity: schizophrenia and schizoaffective disorder
* neurological comorbidity: recent cerebrovascular accident (Less than one month), Parkinson's disease, dementia
* treatment with ketamine received in the four weeks preceding the inclusion
* impaired judgment, cognitive or massive sensory impairment not allowing to receive clear information
* oral antidepressant treatment introduced less than four weeks ago
* dosage of oral antidepressant treatment upper than the marketing authorization for more than four weeks
* patient not covered by the social security system
* refusal to sign the consent
* minor patient or guardianship
* pregnant women (implementation of a urine pregnancy test before inclusion for women of childbearing age)
* lactating women
* intolerance or allergic reaction to ketamine or milnacipran.
* contraindications to the association of ketamine or milnacipran with the patient's usual treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
MADRS Score | At day 1, At day 2
  Measure of the change of Depression Intensity

SECONDARY OUTCOMES:
EUROHIS-QOL 8 | at day 0, at day 15
  Measure of the improvement of quality of life after 15 days of treatment. EUROHIS-QOL 8-item index, a shortened version of the World Health Organization Quality of Life Instrument-Abbreviated Version (WHOQOL-BREF).
Number of request of early death (suicidal intentions or euthanasia or physician-assisted suicide) | at day 0, at day 1, at day 2, at day 4, at day 8, at day 15
  measure request of suicidal intentions made by the patient on explicit request of the clinician.
Hospital Anxiety and Depression scale (HAD) | at day 0, at day 1, at day 2, at day 4, at day 8, at day 15
  The items of the scale limit confounding factors related to physical comorbidity . The answers are simple and quick . It is a wide choice and recommended for depression studies in palliative care.
MADRS Score | at day 0, at day 4, at day 8, at day 15
  The MADRS scale quantifies the intensity of depressive symptoms, determine the number of responders (reduction in the initial score greater than or equal to 50%) and the number of patients in remission (score less than 7).
Clinical Global Impression (CGI) Score | at day 0, at day 1, at day 2, at day 4, at day 8, at day 15
  These hetero fast and well validated assessments help to complete the assessment by the clinician on the severity of the patient's situation and overall improvement
Global Assessment Scale Operation (EGF) | at day 0, at day 15
  Global Assessment of Functioning is a numerical scale ( from 0 to 100) used to evaluate the psychological, social and work of an individual .
Edmonton Symptom Assessment System ( ESAS ) | at day 0, at day 1, at day 2, at day 4, at day 8, at day 15
  Symptom Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Antoine LEMAIRE, MD, Study Chair — Hospital of Valenciennes
Locations (9):
- France (9):
  - Chu Amiens Picardie, Amiens
  - Ch Calais, Calais
  - Maison Medicale Jean Xxiii - Lille, Lille
  - University Hospital,, Lille
  - Groupt Hopitaux Instit Catho de Lille - Lomme, Lomme
  - C.H de Roubaix, Roubaix
  - Ch Ghpso Senlis, Senlis
  - Ch Tourcoing, Tourcoing
  - Centre Hospitalier de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- [Background] Temel JS, Greer JA, Admane S, Gallagher ER, Jackson VA, Lynch TJ, Lennes IT, Dahlin CM, Pirl WF. Longitudinal perceptions of prognosis and goals of therapy in patients with metastatic non-small-cell lung cancer: results of a randomized study of early palliative care. J Clin Oncol. 2011 Jun 10;29(17):2319-26. doi: 10.1200/JCO.2010.32.4459. Epub 2011 May 9. PMID 21555700
- [Background] Lepine JP, Gasquet I, Kovess V, Arbabzadeh-Bouchez S, Negre-Pages L, Nachbaur G, Gaudin AF. [Prevalence and comorbidity of psychiatric disorders in the French general population]. Encephale. 2005 Mar-Apr;31(2):182-94. doi: 10.1016/s0013-7006(05)82385-1. French. PMID 15959445
- [Background] Mitchell AJ, Chan M, Bhatti H, Halton M, Grassi L, Johansen C, Meader N. Prevalence of depression, anxiety, and adjustment disorder in oncological, haematological, and palliative-care settings: a meta-analysis of 94 interview-based studies. Lancet Oncol. 2011 Feb;12(2):160-74. doi: 10.1016/S1470-2045(11)70002-X. Epub 2011 Jan 19. PMID 21251875
- [Background] Atassi N, Cook A, Pineda CM, Yerramilli-Rao P, Pulley D, Cudkowicz M. Depression in amyotrophic lateral sclerosis. Amyotroph Lateral Scler. 2011 Mar;12(2):109-12. doi: 10.3109/17482968.2010.536839. Epub 2010 Nov 24. PMID 21091399
- [Background] Rutledge T, Reis VA, Linke SE, Greenberg BH, Mills PJ. Depression in heart failure a meta-analytic review of prevalence, intervention effects, and associations with clinical outcomes. J Am Coll Cardiol. 2006 Oct 17;48(8):1527-37. doi: 10.1016/j.jacc.2006.06.055. Epub 2006 Sep 26. PMID 17045884
- [Background] Araujo SM, de Bruin VM, Daher Ede F, Almeida GH, Medeiros CA, de Bruin PF. Risk factors for depressive symptoms in a large population on chronic hemodialysis. Int Urol Nephrol. 2012 Aug;44(4):1229-35. doi: 10.1007/s11255-011-0032-9. Epub 2011 Jul 22. PMID 21779919
- [Background] Koenig HG, George LK, Peterson BL, Pieper CF. Depression in medically ill hospitalized older adults: prevalence, characteristics, and course of symptoms according to six diagnostic schemes. Am J Psychiatry. 1997 Oct;154(10):1376-83. doi: 10.1176/ajp.154.10.1376. PMID 9326819
- [Background] Lloyd-Williams M, Friedman T, Rudd N. A survey of antidepressant prescribing in the terminally ill. Palliat Med. 1999 May;13(3):243-8. doi: 10.1191/026921699676753309. PMID 10474711
- [Background] Goldberg RJ, Mor V. A survey of psychotropic use in terminal cancer patients. Psychosomatics. 1985 Sep;26(9):745-8, 751. doi: 10.1016/S0033-3182(85)72803-4. No abstract available. PMID 4048377
- [Background] Rumsfeld JS, Havranek E, Masoudi FA, Peterson ED, Jones P, Tooley JF, Krumholz HM, Spertus JA; Cardiovascular Outcomes Research Consortium. Depressive symptoms are the strongest predictors of short-term declines in health status in patients with heart failure. J Am Coll Cardiol. 2003 Nov 19;42(10):1811-7. doi: 10.1016/j.jacc.2003.07.013. PMID 14642693
- [Background] Cubo E, Bernard B, Leurgans S, Raman R. Cognitive and motor function in patients with Parkinson's disease with and without depression. Clin Neuropharmacol. 2000 Nov-Dec;23(6):331-4. doi: 10.1097/00002826-200011000-00006. PMID 11575867
- [Background] Lyketsos CG, Steele C, Baker L, Galik E, Kopunek S, Steinberg M, Warren A. Major and minor depression in Alzheimer's disease: prevalence and impact. J Neuropsychiatry Clin Neurosci. 1997 Fall;9(4):556-61. doi: 10.1176/jnp.9.4.556. PMID 9447496
- [Background] Aimonino N, Tibaldi V, Barale S, Bardelli B, Pilon S, Marchetto C, Zanocchi M, Molaschi M. Depressive symptoms and quality of life in elderly patients with exacerbation of chronic obstructive pulmonary disease or cardiac heart failure: preliminary data of a randomized controlled trial. Arch Gerontol Geriatr. 2007;44 Suppl 1:7-12. doi: 10.1016/j.archger.2007.01.002. PMID 17317428
- [Background] Newport DJ, Nemeroff CB. Assessment and treatment of depression in the cancer patient. J Psychosom Res. 1998 Sep;45(3):215-37. doi: 10.1016/s0022-3999(98)00011-7. PMID 9776368
- [Background] Rhondali W, Perceau E, Berthiller J, Saltel P, Trillet-Lenoir V, Tredan O, Coulon JP, Bruera E, Filbet M. Frequency of depression among oncology outpatients and association with other symptoms. Support Care Cancer. 2012 Nov;20(11):2795-802. doi: 10.1007/s00520-012-1401-3. Epub 2012 Feb 17. PMID 22350596
- [Background] Onitilo AA, Nietert PJ, Egede LE. Effect of depression on all-cause mortality in adults with cancer and differential effects by cancer site. Gen Hosp Psychiatry. 2006 Sep-Oct;28(5):396-402. doi: 10.1016/j.genhosppsych.2006.05.006. PMID 16950374
- [Background] Satin JR, Linden W, Phillips MJ. Depression as a predictor of disease progression and mortality in cancer patients: a meta-analysis. Cancer. 2009 Nov 15;115(22):5349-61. doi: 10.1002/cncr.24561. PMID 19753617
- [Background] Lloyd-Williams M, Shiels C, Taylor F, Dennis M. Depression--an independent predictor of early death in patients with advanced cancer. J Affect Disord. 2009 Feb;113(1-2):127-32. doi: 10.1016/j.jad.2008.04.002. Epub 2008 Jun 16. PMID 18558439
- [Background] DiMatteo MR, Lepper HS, Croghan TW. Depression is a risk factor for noncompliance with medical treatment: meta-analysis of the effects of anxiety and depression on patient adherence. Arch Intern Med. 2000 Jul 24;160(14):2101-7. doi: 10.1001/archinte.160.14.2101. PMID 10904452
- [Background] Blank K, Robison J, Doherty E, Prigerson H, Duffy J, Schwartz HI. Life-sustaining treatment and assisted death choices in depressed older patients. J Am Geriatr Soc. 2001 Feb;49(2):153-61. doi: 10.1046/j.1532-5415.2001.49036.x. PMID 11207869
- [Background] Rosenfeld KE, Wenger NS, Phillips RS, Connors AF, Dawson NV, Layde P, Califf RM, Liu H, Lynn J, Oye RK. Factors associated with change in resuscitation preference of seriously ill patients. The SUPPORT Investigators. Study to Understand Prognoses and Preferences for Outcomes and Risks of Treatments. Arch Intern Med. 1996 Jul 22;156(14):1558-64. PMID 8687264
- [Background] Breitbart W, Rosenfeld B, Pessin H, Kaim M, Funesti-Esch J, Galietta M, Nelson CJ, Brescia R. Depression, hopelessness, and desire for hastened death in terminally ill patients with cancer. JAMA. 2000 Dec 13;284(22):2907-11. doi: 10.1001/jama.284.22.2907. PMID 11147988
- [Background] Haverkate I, Onwuteaka-Philipsen BD, van Der Heide A, Kostense PJ, van Der Wal G, van Der Maas PJ. Refused and granted requests for euthanasia and assisted suicide in the Netherlands: interview study with structured questionnaire. BMJ. 2000 Oct 7;321(7265):865-6. doi: 10.1136/bmj.321.7265.865. No abstract available. PMID 11021864
- [Background] Meier DE, Emmons CA, Litke A, Wallenstein S, Morrison RS. Characteristics of patients requesting and receiving physician-assisted death. Arch Intern Med. 2003 Jul 14;163(13):1537-42. doi: 10.1001/archinte.163.13.1537. PMID 12860575
- [Background] Buiting HM, Gevers JK, Rietjens JA, Onwuteaka-Philipsen BD, van der Maas PJ, van der Heide A, van Delden JJ. Dutch criteria of due care for physician-assisted dying in medical practice: a physician perspective. J Med Ethics. 2008 Sep;34(9):e12. doi: 10.1136/jme.2008.024976. PMID 18757612
- [Background] Rietjens JA, van der Maas PJ, Onwuteaka-Philipsen BD, van Delden JJ, van der Heide A. Two Decades of Research on Euthanasia from the Netherlands. What Have We Learnt and What Questions Remain? J Bioeth Inq. 2009 Sep;6(3):271-283. doi: 10.1007/s11673-009-9172-3. Epub 2009 Jul 28. PMID 19718271
- [Background] Emanuel LL. Facing requests for physician-assisted suicide: toward a practical and principled clinical skill set. JAMA. 1998 Aug 19;280(7):643-7. doi: 10.1001/jama.280.7.643. PMID 9718058
- [Background] Rayner L, Price A, Hotopf M, Higginson IJ. The development of evidence-based European guidelines on the management of depression in palliative cancer care. Eur J Cancer. 2011 Mar;47(5):702-12. doi: 10.1016/j.ejca.2010.11.027. Epub 2011 Jan 4. PMID 21211961
- [Background] Rayner L, Price A, Evans A, Valsraj K, Hotopf M, Higginson IJ. Antidepressants for the treatment of depression in palliative care: systematic review and meta-analysis. Palliat Med. 2011 Jan;25(1):36-51. doi: 10.1177/0269216310380764. Epub 2010 Oct 8. PMID 20935027
- [Background] Ujeyl M, Muller-Oerlinghausen B. [Antidepressants for treatment of depression in palliative patients : a systematic literature review]. Schmerz. 2012 Sep;26(5):523-36. doi: 10.1007/s00482-012-1221-x. German. PMID 22968366
- [Background] Willner P, Scheel-Kruger J, Belzung C. The neurobiology of depression and antidepressant action. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 1):2331-71. doi: 10.1016/j.neubiorev.2012.12.007. Epub 2012 Dec 19. PMID 23261405
- [Background] Mion G, Villevieille T. Ketamine pharmacology: an update (pharmacodynamics and molecular aspects, recent findings). CNS Neurosci Ther. 2013 Jun;19(6):370-80. doi: 10.1111/cns.12099. Epub 2013 Apr 10. PMID 23575437
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Li N, Lee B, Liu RJ, Banasr M, Dwyer JM, Iwata M, Li XY, Aghajanian G, Duman RS. mTOR-dependent synapse formation underlies the rapid antidepressant effects of NMDA antagonists. Science. 2010 Aug 20;329(5994):959-64. doi: 10.1126/science.1190287. PMID 20724638
- [Background] Li N, Liu RJ, Dwyer JM, Banasr M, Lee B, Son H, Li XY, Aghajanian G, Duman RS. Glutamate N-methyl-D-aspartate receptor antagonists rapidly reverse behavioral and synaptic deficits caused by chronic stress exposure. Biol Psychiatry. 2011 Apr 15;69(8):754-61. doi: 10.1016/j.biopsych.2010.12.015. Epub 2011 Feb 3. PMID 21292242
- [Background] Monteggia LM, Gideons E, Kavalali ET. The role of eukaryotic elongation factor 2 kinase in rapid antidepressant action of ketamine. Biol Psychiatry. 2013 Jun 15;73(12):1199-203. doi: 10.1016/j.biopsych.2012.09.006. Epub 2012 Oct 11. PMID 23062356
- [Background] Beurel E, Song L, Jope RS. Inhibition of glycogen synthase kinase-3 is necessary for the rapid antidepressant effect of ketamine in mice. Mol Psychiatry. 2011 Nov;16(11):1068-70. doi: 10.1038/mp.2011.47. Epub 2011 Apr 19. No abstract available. PMID 21502951
- [Background] Li X, Jope RS. Is glycogen synthase kinase-3 a central modulator in mood regulation? Neuropsychopharmacology. 2010 Oct;35(11):2143-54. doi: 10.1038/npp.2010.105. Epub 2010 Jul 28. PMID 20668436
- [Background] Akinfiresoye L, Tizabi Y. Antidepressant effects of AMPA and ketamine combination: role of hippocampal BDNF, synapsin, and mTOR. Psychopharmacology (Berl). 2013 Nov;230(2):291-8. doi: 10.1007/s00213-013-3153-2. Epub 2013 Jun 4. PMID 23732839
- [Background] Autry AE, Adachi M, Nosyreva E, Na ES, Los MF, Cheng PF, Kavalali ET, Monteggia LM. NMDA receptor blockade at rest triggers rapid behavioural antidepressant responses. Nature. 2011 Jun 15;475(7354):91-5. doi: 10.1038/nature10130. PMID 21677641
- [Background] Koike H, Iijima M, Chaki S. Involvement of AMPA receptor in both the rapid and sustained antidepressant-like effects of ketamine in animal models of depression. Behav Brain Res. 2011 Oct 10;224(1):107-11. doi: 10.1016/j.bbr.2011.05.035. Epub 2011 Jun 6. PMID 21669235
- [Background] Rasmussen KG, Lineberry TW, Galardy CW, Kung S, Lapid MI, Palmer BA, Ritter MJ, Schak KM, Sola CL, Hanson AJ, Frye MA. Serial infusions of low-dose ketamine for major depression. J Psychopharmacol. 2013 May;27(5):444-50. doi: 10.1177/0269881113478283. Epub 2013 Feb 20. PMID 23428794
- [Background] Price RB, Nock MK, Charney DS, Mathew SJ. Effects of intravenous ketamine on explicit and implicit measures of suicidality in treatment-resistant depression. Biol Psychiatry. 2009 Sep 1;66(5):522-6. doi: 10.1016/j.biopsych.2009.04.029. Epub 2009 Jul 9. PMID 19545857
- [Background] Thakurta RG, Das R, Bhattacharya AK, Saha D, Sen S, Singh OP, Bisui B. Rapid response with ketamine on suicidal cognition in resistant depression. Indian J Psychol Med. 2012 Apr;34(2):170-5. doi: 10.4103/0253-7176.101793. PMID 23162195
- [Background] Glue P, Gulati A, Le Nedelec M, Duffull S. Dose- and exposure-response to ketamine in depression. Biol Psychiatry. 2011 Aug 15;70(4):e9-10; author reply e11-2. doi: 10.1016/j.biopsych.2010.11.031. Epub 2011 Apr 8. No abstract available. PMID 21481846
- [Background] Loo CK, Katalinic N, Garfield JB, Sainsbury K, Hadzi-Pavlovic D, Mac-Pherson R. Neuropsychological and mood effects of ketamine in electroconvulsive therapy: a randomised controlled trial. J Affect Disord. 2012 Dec 15;142(1-3):233-40. doi: 10.1016/j.jad.2012.04.032. Epub 2012 Aug 2. PMID 22858219
- [Background] Thakurta RG, Ray P, Kanji D, Das R, Bisui B, Singh OP. Rapid Antidepressant Response with Ketamine: Is it the Solution to Resistant Depression? Indian J Psychol Med. 2012 Jan;34(1):56-60. doi: 10.4103/0253-7176.96161. PMID 22661809
- [Background] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Background] Cusin C, Hilton GQ, Nierenberg AA, Fava M. Long-term maintenance with intramuscular ketamine for treatment-resistant bipolar II depression. Am J Psychiatry. 2012 Aug;169(8):868-9. doi: 10.1176/appi.ajp.2012.12020219. No abstract available. PMID 22854933
- [Background] Paslakis G, Gilles M, Meyer-Lindenberg A, Deuschle M. Oral administration of the NMDA receptor antagonist S-ketamine as add-on therapy of depression: a case series. Pharmacopsychiatry. 2010 Jan;43(1):33-5. doi: 10.1055/s-0029-1237375. Epub 2009 Dec 11. No abstract available. PMID 20013614
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710